CLINICAL TRIAL: NCT03086499
Title: Clustering Among the Clinical Profiles of Patients With Pectus Excavatum
Acronym: PECTUS-cluster
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0094
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Funnel Chest
Keywords: pectus excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: Patients with pectus excavatum having consulted at the Montpellier University Hospital and who have had corrective surgery.

SUMMARY:
The primary objective of this study is to describe the relative distances between patient clinical profiles (i.e. patient clustering) in multivariate space.

DETAILED DESCRIPTION:
Observational data will be collected from patient files and submitted to clustering analyses. Then clusters will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with pectus excavatum
* The patient has had corrective surgery

Exclusion Criteria:

* The patient has expressed opposition to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pectus excavatum having consulted at the Montpellier University Hospital and who have had corrective surgery.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
The number of clusters found | Day 0 (transversal, retrospective study)
  The number of clusters found among clinical profiles

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe Berthet, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- See also: PECTUS-cluster on the Open Science Framework — http://osf.io/f2jue